CLINICAL TRIAL: NCT04394585
Title: A Study Evaluating Effect of Smart Phone App-based Human Coaching Program on QOL in Patients Who Underwent Gastrectomy for Stage I Gastric Cancer
Brief Title: Effect of Smart Phone App-based Human Coaching Program in Gastrectomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Bang Wool Eom, Dr, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1910242
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Stage I Gastric Cancer
Keywords: gastric cancer; quality of life; smart phone app; human coaching program
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smart phone app group (Experimental): Patients used smart phone app based human coaching program for 3 months postoperatively.
  Interventions: Behavioral: smart phone app based human coaching program
- Nutritional consultation group (Active Comparator): Patients have two consulting with clinical nutritionist at 1 month and 3 months postoperatively.
  Interventions: Behavioral: smart phone app based human coaching program

INTERVENTIONS:
Behavioral: smart phone app based human coaching program — 1. experimental arm
     * 1:1 coaching using smart phone app
     * Patients are provided several articles about postoperative care (symptom management, diet, and exercise) in the app.
     * Patients are encouraged to report their diet diaries and exercise everyday by the coach.
     * Patients can ask to the coach using the app and the coach answer when they check them.
  2. Comparator arm - Patient have consulting with clinical nutritionist at 1 month and 3 months postoperatively.

SUMMARY:
This study is a single center, prospective, randomized controlled study. The aim of this study is to evaluate the effect of smart phone app-based human coaching program on QOL in patients who underwent gastrectomy for stage I gastric cancer. The hypothesis of this study is the patients who used smart phone app-based human coaching program for three months after surgery will have better QOL than patients who did not use it. The QOL will be assessed using EORTC QLQ C30 and STO22 at 3 months postoperatively. The secondary endpoints are QOL at 6 months postoperatively, 12 months postoperative, food intake, body composition, and nutritional indicators from blood test.

DETAILED DESCRIPTION:
< Patient enrollment>

* 90 patients in each group, a total of 180 patients
* 1:1 Randomization using permutated mixed block randomization
* stratified by surgical extent (distal gastrectomy vs. total gastrectomy)
* using nQuery program and web-based management system
* Before discharge, patients are informed how to use the smart phone app and registered to the app.
* Patients use the app after discharge until 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 19 or more
* patient diagnosed as stage I in preoperative examination
* planned distal gastrectomy or total gastrectomy
* patient who can use smart phone app or whose family can help the
* patient to use the smart phone app

Exclusion Criteria:

* pregnant
* disabled to communication
* patient who cannot use smart phone app

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eating restriction score (XEatR) at 1 month postoperatively | 1 month postoperatively
  Eating resection scale is calculated according to the following equation. a. Add questionnaire items 41,42, 43 and 46 and divide this sum by the number of items (4): EatR = (Q41+Q42+Q43+Q46)/4 b. Carry out a linear transformation to convert to a 1-100 scale: XEatR = (EatR-1)*100/3 The 4 items are belong to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) STO22. Each item has a value among 1, 2, 3, and 4 according to the answer and the scale score has a value ranging 0 (minimum) to 100 (maximum). Higher scores mean having more symptom and worse quality of life.
Eating restriction score (XEatR) at 3 months postoperatively | 3 months postoperatively
  Eating resection scale is calcuated according to the following equation.
  1. Add questionnaire items 41,42, 43 and 46 and divide this sum by the number of items (4):
     EatR = (Q41+Q42+Q43+Q46)/4
  2. Carry out a linear transformation to convert to a 1-100 scale:
  XEatR = (EatR-1)*100/3
  The 4 items are belong to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) STO22.
  Each item has a value among 1, 2, 3, and 4 according to the answer and the scale score has a value ranging 0 (minimum) to 100 (maximum).
  Higher scores mean having more symptom and worse quality of life.

SECONDARY OUTCOMES:
Eating restriction score (XEatR) at 6 months postoperatively | 6 months postoperatively
  Eating resection scale is calcuated according to the following equation.
  1. Add questionnaire items 41,42, 43 and 46 and divide this sum by the number of items (4):
     EatR = (Q41+Q42+Q43+Q46)/4
  2. Carry out a linear transformation to convert to a 1-100 scale:
  XEatR = (EatR-1)*100/3
  The 4 items are belong to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) STO22.
  Each item has a value among 1, 2, 3, and 4 according to the answer and the scale score has a value ranging 0 (minimum) to 100 (maximum).
  Higher scores mean having more symptom and worse quality of life.
Eating restriction score (XEatR) at 12 months postoperatively | 12 months postoperatively
  Eating resection scale is calcuated according to the following equation.
  1. Add questionnaire items 41,42, 43 and 46 and divide this sum by the number of items (4):
     EatR = (Q41+Q42+Q43+Q46)/4
  2. Carry out a linear transformation to convert to a 1-100 scale:
  XEatR = (EatR-1)*100/3
  The 4 items are belong to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) STO22.
  Each item has a value among 1, 2, 3, and 4 according to the answer and the scale score has a value ranging 0 (minimum) to 100 (maximum).
  Higher scores mean having more symptom and worse quality of life.
food intake | discharge day: up to 3 weeks postoperatively,1 month postoperatively
  difference of food amount between discharge day and postoperative 1 month
Body weight | 3 months postoperatively
  patient's weight in kilograms
serum albumin | 3 months postoperatively
  g/dL
serum protein | 3 months postoperatively
  g/dL
serum cholesterol | 3 months postoperatively
  g/dL
seum hemoglobin | 3 months postoperatively
  g/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Bang Wool Eom, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eom BW, Han M, Yoon HM, Kim YW, Kim SY, Oh JM, Wie GA, Ryu KW. Improvement in Quality of Life After Early Interactive Human Coaching via a Mobile App in Postgastrectomy Patients With Gastric Cancer: Prospective Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Dec 18;13:e75445. doi: 10.2196/75445. PMID 41411643
- [Derived] Kim HJ, Yoon HM, Ryu KW, Kim YW, Kim SY, Oh JM, Wie GA, Ko H, Lee J, Kim Y, Cho H, Eom BW. An early interactive human coaching via a mobile application to improve quality of life in patients who underwent gastrectomy for gastric cancer: Design and protocol of a randomized controlled trial. PLoS One. 2022 Dec 9;17(12):e0278370. doi: 10.1371/journal.pone.0278370. eCollection 2022. PMID 36490244